CLINICAL TRIAL: NCT01451697
Title: Cognitive Remediation for Neuropsychological Impairment in Compulsive Hoarding
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIMA003472HI
Record Dates: First submitted 2011-10-10; First posted 2011-10-14 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Hoarding Disorder; Attentional Impairment
MeSH Terms: conditions — Hoarding Disorder | interventions — Cognitive Remediation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Cognitive Remediation (Experimental): The remediation intervention will consist of a sequence of computerized cognitive exercises designed to improve a variety of aspects of attention, through repeated drill-and-practice (Bell, Bryson, Greig, Corcoran, & Wexler, 2001; Bracy, 1995; Kurtz et al., 2007). Exercises will be started and continued at the highest level of difficulty, in order to best establish improvement over time. Components of the planned intervention produce performance gains on practiced tasks (e.g., Wexler et al., 1997) and generalization of improvement to other tasks (Kurtz et al., 2007). All training on computer exercises will be conducted with coaching from staff trained in these procedures.
  Interventions: Behavioral: Cognitive Remediation
- Control (Placebo) (Placebo Comparator): The placebo control condition will consist of structured relaxation training, which will involve viewing and participating with meditation and stress-reduction DVDs, and listening to and following a CD of Progressive Muscle Relaxation. Participants will benefit from learning stress reduction techniques in this condition, but will not exercise any of the cognitive domains of interest targeted in the treatment group.
  Interventions: Behavioral: Control (Placebo)

INTERVENTIONS:
Behavioral: Cognitive Remediation — A computerized cognitive remediation program focused on attentional training will be used.
  Arms: Experimental: Cognitive Remediation
Behavioral: Control (Placebo) — The control condition will involve relaxation training.
  Arms: Control (Placebo)

SUMMARY:
The primary aim of this pilot randomized controlled trial is to examine whether cognitive remediation, compared to a placebo, improves attention and related cognitive functions in patients with compulsive hoarding. The primary hypothesis is that compulsive hoarding patients who are treated with cognitive remediation will demonstrate improved cognitive skills at post-treatment compared to patients receiving placebo. This will be especially true of attention; memory and executive function skills may also be improved.

DETAILED DESCRIPTION:
The primary aim of this pilot randomized controlled trial is to examine whether cognitive remediation, compared to a placebo, improves attention and related cognitive functions in patients with compulsive hoarding. Previous research has demonstrated that hoarders have diminished neuropsychological abilities, particularly in the areas of attention, memory, and executive function; and that cognitive remediation improves those functions in populations that are similarly impaired, such as in individuals with schizophrenia. The investigators will thus randomize 20 patients with compulsive hoarding to receive either cognitive remediation or a placebo condition. Before and after treatment, the investigators aim to assess the effects of cognitive remediation on neuropsychological functioning and hoarding severity. The primary specific aim is to examine whether cognitive remediation improves cognitive function in compulsive hoarders. The investigators hypothesize that compulsive hoarding patients who are treated with cognitive remediation will demonstrate improved cognitive skills at post-treatment compared to patients receiving placebo. This will be especially true of attention; memory and executive function skills may also be improved. A secondary, exploratory aim is to examine whether cognitive remediation improves hoarding severity, compared to placebo. The ultimate goal of this research is to determine the feasibility and appropriateness of pursuing larger-scale studies of the promising new approach of combining cognitive remediation with other treatments for compulsive hoarding-particularly cognitive-behavioral therapy (CBT).

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years of age,
* have a current primary diagnosis of hoarding disorder
* have no untreated and/or unstable concurrent psychiatric diagnoses
* have a score on the ADHDSS that is one standard deviation or more above the mean
* have an Attentional Composite score on the computerized battery of neuropsychological tests (Doniger, 2010) that is one standard deviation or more below the mean
* be stable on all psychotropic medications during and up to four weeks preceding enrollment in the study

Exclusion Criteria:

* currently taking any cognitive enhancers or stimulants
* people with a history of Multiple Sclerosis, Traumatic Brain Injury, loss of consciousness lasting more than 5 minutes, seizures, dementia, or other organic brain-related disorders
* current Alcohol or Substance Abuse and/or a history of Alcohol or Substance Dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Continuous Performance Task (computerized version): change from Baseline in Attentional Functioning at 8 Weeks | Week 0 (Baseline) and Week 8 (Endpoint)
  This measure is a computerized assessment of attention, memory, and executive functioning. The investigators will use this measure to assess change in those cognitive domains between Baseline (Week 0) and Endpoint (Week 8).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer DiMauro, BA, Principal Investigator — Hartford Hospital; David F Tolin, PhD, Study Director — Hartford Hospital
Locations (1):
- Anxiety Disorders Center, Institute of Living/Hartford, Hartford, Connecticut, United States

REFERENCES:
- [Background] Abramowitz JS, Wheaton MG, Storch EA. The status of hoarding as a symptom of obsessive-compulsive disorder. Behav Res Ther. 2008 Sep;46(9):1026-33. doi: 10.1016/j.brat.2008.05.006. Epub 2008 Jun 27. PMID 18684434
- [Background] Auriel E, Hausdorff JM, Herman T, Simon ES, Giladi N. Effects of methylphenidate on cognitive function and gait in patients with Parkinson's disease: a pilot study. Clin Neuropharmacol. 2006 Jan-Feb;29(1):15-7. doi: 10.1097/00002826-200601000-00005. PMID 16518128
- [Background] Barbieri L, Boggian I, Falloon I, Lamonaca D; Centro Diurno 5 (CD5) collaborators. Problem-solving skills for cognitive rehabilitation among persons with chronic psychotic disorders in Italy. Psychiatr Serv. 2006 Feb;57(2):172-4. doi: 10.1176/appi.ps.57.2.172. PMID 16452691
- [Background] BECK LH, BRANSOME ED Jr, MIRSKY AF, ROSVOLD HE, SARASON I. A continuous performance test of brain damage. J Consult Psychol. 1956 Oct;20(5):343-50. doi: 10.1037/h0043220. No abstract available. PMID 13367264
- [Background] Beck AT, Beck RW. Screening depressed patients in family practice. A rapid technic. Postgrad Med. 1972 Dec;52(6):81-5. doi: 10.1080/00325481.1972.11713319. No abstract available. PMID 4635613
- [Background] Bell M, Bryson G, Greig T, Corcoran C, Wexler BE. Neurocognitive enhancement therapy with work therapy: effects on neuropsychological test performance. Arch Gen Psychiatry. 2001 Aug;58(8):763-8. doi: 10.1001/archpsyc.58.8.763. PMID 11483142
- [Background] Bernal G, Bonilla J, Padilla-Cotto L, Perez-Prado EM. Factors associated to outcome in psychotherapy: an effectiveness study in Puerto Rico. J Clin Psychol. 1998 Apr;54(3):329-42. doi: 10.1002/(sici)1097-4679(199804)54:33.0.co;2-k. PMID 9545170
- [Background] Castellanos FX, Sonuga-Barke EJ, Milham MP, Tannock R. Characterizing cognition in ADHD: beyond executive dysfunction. Trends Cogn Sci. 2006 Mar;10(3):117-23. doi: 10.1016/j.tics.2006.01.011. Epub 2006 Feb 7. PMID 16460990
- [Background] Diefenbach GJ, Abramowitz JS, Norberg MM, Tolin DF. Changes in quality of life following cognitive-behavioral therapy for obsessive-compulsive disorder. Behav Res Ther. 2007 Dec;45(12):3060-8. doi: 10.1016/j.brat.2007.04.014. Epub 2007 May 10. PMID 17559803
- [Background] Dwolatzky T, Whitehead V, Doniger GM, Simon ES, Schweiger A, Jaffe D, Chertkow H. Validity of a novel computerized cognitive battery for mild cognitive impairment. BMC Geriatr. 2003 Nov 2;3:4. doi: 10.1186/1471-2318-3-4. PMID 14594456
- [Background] Elstein D, Guedalia J, Doniger GM, Simon ES, Antebi V, Arnon Y, Zimran A. Computerized cognitive testing in patients with type I Gaucher disease: effects of enzyme replacement and substrate reduction. Genet Med. 2005 Feb;7(2):124-30. doi: 10.1097/01.gim.0000153666.23707.ba. PMID 15714080
- [Background] Endicott J, Nee J, Harrison W, Blumenthal R. Quality of Life Enjoyment and Satisfaction Questionnaire: a new measure. Psychopharmacol Bull. 1993;29(2):321-6. PMID 8290681
- [Background] Epstein JN, Johnson DE, Varia IM, Conners CK. Neuropsychological assessment of response inhibition in adults with ADHD. J Clin Exp Neuropsychol. 2001 Jun;23(3):362-71. doi: 10.1076/jcen.23.3.362.1186. PMID 11404813
- [Background] Frost RO, Gross RC. The hoarding of possessions. Behav Res Ther. 1993 May;31(4):367-81. doi: 10.1016/0005-7967(93)90094-b. PMID 8512538
- [Background] Frost RO, Hartl TL. A cognitive-behavioral model of compulsive hoarding. Behav Res Ther. 1996 Apr;34(4):341-50. doi: 10.1016/0005-7967(95)00071-2. PMID 8871366
- [Background] Frost RO, Kim HJ, Morris C, Bloss C, Murray-Close M, Steketee G. Hoarding, compulsive buying and reasons for saving. Behav Res Ther. 1998 Jul-Aug;36(7-8):657-64. doi: 10.1016/s0005-7967(98)00056-4. PMID 9682522
- [Background] Frost RO, Krause MS, Steketee G. Hoarding and obsessive-compulsive symptoms. Behav Modif. 1996 Jan;20(1):116-32. doi: 10.1177/01454455960201006. PMID 8561769
- [Background] Frost RO, Steketee G, Grisham J. Measurement of compulsive hoarding: saving inventory-revised. Behav Res Ther. 2004 Oct;42(10):1163-82. doi: 10.1016/j.brat.2003.07.006. PMID 15350856
- [Background] Galbiati S, Recla M, Pastore V, Liscio M, Bardoni A, Castelli E, Strazzer S. Attention remediation following traumatic brain injury in childhood and adolescence. Neuropsychology. 2009 Jan;23(1):40-9. doi: 10.1037/a0013409. PMID 19210031
- [Background] Grisham JR, Brown TA, Liverant GI, Campbell-Sills L. The distinctiveness of compulsive hoarding from obsessive-compulsive disorder. J Anxiety Disord. 2005;19(7):767-79. doi: 10.1016/j.janxdis.2004.09.003. PMID 16076423
- [Background] Grisham JR, Brown TA, Savage CR, Steketee G, Barlow DH. Neuropsychological impairment associated with compulsive hoarding. Behav Res Ther. 2007 Jul;45(7):1471-83. doi: 10.1016/j.brat.2006.12.008. Epub 2007 Jan 12. PMID 17341416
- [Background] Hartl TL, Duffany SR, Allen GJ, Steketee G, Frost RO. Relationships among compulsive hoarding, trauma, and attention-deficit/hyperactivity disorder. Behav Res Ther. 2005 Feb;43(2):269-76. doi: 10.1016/j.brat.2004.02.002. PMID 15629755
- [Background] Hartl TL, Frost RO, Allen GJ, Deckersbach T, Steketee G, Duffany SR, Savage CR. Actual and perceived memory deficits in individuals with compulsive hoarding. Depress Anxiety. 2004;20(2):59-69. doi: 10.1002/da.20010. PMID 15390215
- [Background] Iervolino AC, Perroud N, Fullana MA, Guipponi M, Cherkas L, Collier DA, Mataix-Cols D. Prevalence and heritability of compulsive hoarding: a twin study. Am J Psychiatry. 2009 Oct;166(10):1156-61. doi: 10.1176/appi.ajp.2009.08121789. Epub 2009 Aug 17. PMID 19687130
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Kessler RC, Frank RG. The impact of psychiatric disorders on work loss days. Psychol Med. 1997 Jul;27(4):861-73. doi: 10.1017/s0033291797004807. PMID 9234464
- [Background] Kocsis JH, Zisook S, Davidson J, Shelton R, Yonkers K, Hellerstein DJ, Rosenbaum J, Halbreich U. Double-blind comparison of sertraline, imipramine, and placebo in the treatment of dysthymia: psychosocial outcomes. Am J Psychiatry. 1997 Mar;154(3):390-5. doi: 10.1176/ajp.154.3.390. PMID 9054788
- [Background] Kurtz MM, Ragland JD, Bilker W, Gur RC, Gur RE. Comparison of the continuous performance test with and without working memory demands in healthy controls and patients with schizophrenia. Schizophr Res. 2001 Mar 30;48(2-3):307-16. doi: 10.1016/s0920-9964(00)00060-8. PMID 11295383
- [Background] Kurtz MM, Seltzer JC, Shagan DS, Thime WR, Wexler BE. Computer-assisted cognitive remediation in schizophrenia: what is the active ingredient? Schizophr Res. 2007 Jan;89(1-3):251-60. doi: 10.1016/j.schres.2006.09.001. Epub 2006 Oct 27. PMID 17070671
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Leon AC, Shear MK, Portera L, Klerman GL. Assessing impairment in patients with panic disorder: the Sheehan Disability Scale. Soc Psychiatry Psychiatr Epidemiol. 1992 Mar;27(2):78-82. doi: 10.1007/BF00788510. PMID 1594977
- [Background] Lindenmayer JP, McGurk SR, Mueser KT, Khan A, Wance D, Hoffman L, Wolfe R, Xie H. A randomized controlled trial of cognitive remediation among inpatients with persistent mental illness. Psychiatr Serv. 2008 Mar;59(3):241-7. doi: 10.1176/ps.2008.59.3.241. PMID 18308903
- [Background] Medalia A, Aluma M, Tryon W, Merriam AE. Effectiveness of attention training in schizophrenia. Schizophr Bull. 1998;24(1):147-52. doi: 10.1093/oxfordjournals.schbul.a033306. PMID 9502552
- [Background] Medalia A, Dorn H, Watras-Gans S. Treating problem-solving deficits on an acute care psychiatric inpatient unit. Psychiatry Res. 2000 Dec 4;97(1):79-88. doi: 10.1016/s0165-1781(00)00214-6. PMID 11104859
- [Background] Medalia A, Revheim N, Casey M. The remediation of problem-solving skills in schizophrenia. Schizophr Bull. 2001;27(2):259-67. doi: 10.1093/oxfordjournals.schbul.a006872. PMID 11354593
- [Background] Mick E, Faraone SV, Spencer T, Zhang HF, Biederman J. Assessing the validity of the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form in adults with ADHD. J Atten Disord. 2008 Jan;11(4):504-9. doi: 10.1177/1087054707308468. Epub 2007 Oct 12. PMID 17934183
- [Background] O'Connell RG, Bellgrove MA, Dockree PM, Lau A, Fitzgerald M, Robertson IH. Self-Alert Training: volitional modulation of autonomic arousal improves sustained attention. Neuropsychologia. 2008 Apr;46(5):1379-90. doi: 10.1016/j.neuropsychologia.2007.12.018. Epub 2007 Dec 27. PMID 18249419
- [Background] O'Connell RG, Bellgrove MA, Dockree PM, Robertson IH. Cognitive remediation in ADHD: effects of periodic non-contingent alerts on sustained attention to response. Neuropsychol Rehabil. 2006 Dec;16(6):653-65. doi: 10.1080/09602010500200250. PMID 17127571
- [Background] Rohling ML, Faust ME, Beverly B, Demakis G. Effectiveness of cognitive rehabilitation following acquired brain injury: a meta-analytic re-examination of Cicerone et al.'s (2000, 2005) systematic reviews. Neuropsychology. 2009 Jan;23(1):20-39. doi: 10.1037/a0013659. PMID 19210030
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Samuels JF, Bienvenu OJ, Grados MA, Cullen B, Riddle MA, Liang KY, Eaton WW, Nestadt G. Prevalence and correlates of hoarding behavior in a community-based sample. Behav Res Ther. 2008 Jul;46(7):836-44. doi: 10.1016/j.brat.2008.04.004. Epub 2008 Apr 13. PMID 18495084
- [Background] Sartory G, Zorn C, Groetzinger G, Windgassen K. Computerized cognitive remediation improves verbal learning and processing speed in schizophrenia. Schizophr Res. 2005 Jun 15;75(2-3):219-23. doi: 10.1016/j.schres.2004.10.004. Epub 2004 Nov 13. PMID 15885513
- [Background] Steketee G, Frost R. Compulsive hoarding: current status of the research. Clin Psychol Rev. 2003 Dec;23(7):905-27. doi: 10.1016/j.cpr.2003.08.002. PMID 14624821
- [Background] Stevenson CS, Whitmont S, Bornholt L, Livesey D, Stevenson RJ. A cognitive remediation programme for adults with Attention Deficit Hyperactivity Disorder. Aust N Z J Psychiatry. 2002 Oct;36(5):610-6. doi: 10.1046/j.1440-1614.2002.01052.x. PMID 12225443
- [Background] Tolin DF, Frost RO, Steketee G. An open trial of cognitive-behavioral therapy for compulsive hoarding. Behav Res Ther. 2007 Jul;45(7):1461-70. doi: 10.1016/j.brat.2007.01.001. Epub 2007 Jan 16. PMID 17306221
- [Background] Tolin DF, Frost RO, Steketee G, Fitch KE. Family burden of compulsive hoarding: results of an internet survey. Behav Res Ther. 2008 Mar;46(3):334-44. doi: 10.1016/j.brat.2007.12.008. Epub 2008 Jan 3. PMID 18275935
- [Background] Tolin DF, Frost RO, Steketee G, Gray KD, Fitch KE. The economic and social burden of compulsive hoarding. Psychiatry Res. 2008 Aug 15;160(2):200-11. doi: 10.1016/j.psychres.2007.08.008. Epub 2008 Jul 1. PMID 18597855
- [Background] Tolin DF, Kiehl KA, Worhunsky P, Book GA, Maltby N. An exploratory study of the neural mechanisms of decision making in compulsive hoarding. Psychol Med. 2009 Feb;39(2):325-36. doi: 10.1017/S0033291708003371. Epub 2008 May 19. PMID 18485263
- [Background] Tolin DF, Robison JT, Gaztambide S, Blank K. Anxiety disorders in older Puerto Rican primary care patients. Am J Geriatr Psychiatry. 2005 Feb;13(2):150-6. doi: 10.1176/appi.ajgp.13.2.150. PMID 15703324
- [Background] Wagle AC, Berrios GE, Ho L. The cognitive failures questionnaire in psychiatry. Compr Psychiatry. 1999 Nov-Dec;40(6):478-84. doi: 10.1016/s0010-440x(99)90093-7. PMID 10579381
- [Background] Wexler BE, Anderson M, Fulbright RK, Gore JC. Preliminary evidence of improved verbal working memory performance and normalization of task-related frontal lobe activation in schizophrenia following cognitive exercises. Am J Psychiatry. 2000 Oct;157(10):1694-7. doi: 10.1176/appi.ajp.157.10.1694. PMID 11007730
- [Background] Wexler BE, Hawkins KA, Rounsaville B, Anderson M, Sernyak MJ, Green MF. Normal neurocognitive performance after extended practice in patients with schizophrenia. Schizophr Res. 1997 Aug 29;26(2-3):173-80. doi: 10.1016/s0920-9964(97)00053-4. PMID 9323348
- [Background] Woods SP, Lovejoy DW, Ball JD. Neuropsychological characteristics of adults with ADHD: a comprehensive review of initial studies. Clin Neuropsychol. 2002 Feb;16(1):12-34. doi: 10.1076/clin.16.1.12.8336. PMID 11992223
- [Background] Wykes T, Reeder C, Corner J, Williams C, Everitt B. The effects of neurocognitive remediation on executive processing in patients with schizophrenia. Schizophr Bull. 1999;25(2):291-307. doi: 10.1093/oxfordjournals.schbul.a033379. PMID 10416732
- [Background] Wykes T, Reeder C, Williams C, Corner J, Rice C, Everitt B. Are the effects of cognitive remediation therapy (CRT) durable? Results from an exploratory trial in schizophrenia. Schizophr Res. 2003 Jun 1;61(2-3):163-74. doi: 10.1016/s0920-9964(02)00239-6. PMID 12729868